CLINICAL TRIAL: NCT02263352
Title: Systemic Lycopene as an Adjunct to Scaling and Rootplaning in Chronic Periodontitis Patients With Type 2 Diabetes Mellitus
Brief Title: A Clinical Trial to Study the Effect of Lycopene in Patients With Gum Disease and type2 Diabetes Mellitus
Acronym: "SLSRPD"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Collaborators: National Institute of Health and Nutrition (Other Government)
Responsible Party: Principal Investigator, Manasa Ambati, Dr.Manasa Ambati, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/98/12
Record Dates: First submitted 2014-10-01; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Positive Regulation of Oxidative Stress Process
Keywords: Diabetes, Periodontitis, Oxidative stress, Antioxidant
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis | interventions — Weights and Measures; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lycored soft gels , Scaling and Rootplaning. (Experimental): Systemic Lycored soft gels,(Jagsonpal Pharma) was given orally 8mgms/day for 2 months and Scaling and rootplaning (otherwise known as conventional periodontal therapy, non-surgical periodontal therapy, or deep cleaning, is the process of removing or eliminating the etiologic agents - dental plaque, its products, and calculus) which was performed at baseline
  Interventions: Drug: Lycored soft gels Jagsonpal Pharma, Systemic 8mgms/day; Device: Scaling and root planing
- Scaling and Rootplaning only. (Experimental): Scaling and rootplaning(otherwise known as conventional periodontal therapy, non-surgical periodontal therapy, or deep cleaning, is the process of removing or eliminating the etiologic agents - dental plaque, its products, and calculus) which was performed at baseline.
  Interventions: Device: Scaling and root planing

INTERVENTIONS:
Drug: Lycored soft gels Jagsonpal Pharma, Systemic 8mgms/day — Lycopene 8mgms taken orally ,one per day for two months.
  Other Names: rhodopurpurin,non-provitamin A carotenoid,
  Arms: Lycored soft gels , Scaling and Rootplaning.
Device: Scaling and root planing — Scaling and root planing, otherwise known as conventional periodontal therapy, non-surgical periodontal therapy, or deep cleaning, is the process of removing or eliminating the etiologic agents - dental plaque, its products, and calculus
  Other Names: Nonsurgical periodontal therapy, Conventional periodontal therapy.

SUMMARY:
This study was performed to assess the efficacy of systemic lycopene (8 mgms Daily for two months) as an adjunct to scaling and root planing in chronic periodontitis patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This study is a randomized double blinded clinical trial which was performed to assess the efficacy of systemic lycopene (8 mgms Daily for two months) as an adjunct to scaling and root planing in chronic periodontitis patients with type 2 diabetes mellitus. The primary outcome measures were Serum MDA, CRP and Hb1AC. The secondary outcomes were modified gingival index(GI), Probing pocket depth(PPD), and Clinical attachment level(CAL). All the outcomes were measured at baseline, 2 months and 6 months.

The results were that the Lycopene with scaling and root planing group gave:

Statistically significant results in reducing Mean serum MDA levels at 2 months and 6 months respectively.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes

* Patients on oral hypoglycemic drugs with no modification in therapy from the past 12 months
* Chronic periodontitis as per AAP (American Academy of Periodontology) guidelines
* Minimum of 15 natural teeth
* At least four teeth with one or more sites with probing depth (PD) greater than or equal to 5 mm, clinical attachment level (CAL) greater than or equal to 4mm and bleeding on probing (BOP).

Exclusion Criteria:

History of antibiotic therapy within the previous 6 months

* History of anti-inflammatory drugs within the previous 3 months
* Pregnancy and lactation
* Use of contraceptives or any other form of hormone
* Usage of tobacco and tobacco related products
* Periodontal treatment within 12 months.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Serum MDA | 6 Months Post treatment.
  This unique outcome measure was assessed from baseline to 6 months post treatment by spectrophotometric estimation of serum Thiobarbituric acid substances (TBARS). The TBARS Assay measures malondialdehyde (MDA), a reactive compound formed from lipid peroxides that are generated under conditions of oxidative stress. Oxidative modification of lipids occurs with aging and various diseases, and increased oxidative stress is associated with diabetes and its complications. MDA forms an adduct with thiobarbituric acid (TBA). Results are calculated from a standard curve constructed with authentic MDA.

SECONDARY OUTCOMES:
Change in Modified Gingival Index | 6 Months post treatment.
  The change in Modified gingival index from baseline to 6 months post treatment was assessed full mouth at 6 sites /tooth with Hufreidy Periodontal probe.
Change in Probing pocket depth (PPD) | 6 Months post treatment.
  The change in Probing pocket depth from baseline to 6 months post treatment was assessed full mouth at 6 sites /tooth with Hufreidy Periodontal probe.
Change in Clinical attachment level (CAL) | 6 Months post treatment.
  The change in CAL from baseline to 6 months post treatment was assessed full mouth at 6 sites /tooth with Hufreidy Periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Manasa Ambati, MDS(Perio), Principal Investigator — Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre,Road no:5,Kamala nagar,Dilsukhnagar,Hyderabad,India.
Locations (1):
- Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre, Hyderabad, India

REFERENCES:
- [Background] Neyestani TR, Shariatzadeh N, Gharavi A, Kalayi A, Khalaji N. Physiological dose of lycopene suppressed oxidative stress and enhanced serum levels of immunoglobulin M in patients with Type 2 diabetes mellitus: a possible role in the prevention of long-term complications. J Endocrinol Invest. 2007 Nov;30(10):833-8. doi: 10.1007/BF03349224. PMID 18075285
- [Background] Chandra RV, Prabhuji ML, Roopa DA, Ravirajan S, Kishore HC. Efficacy of lycopene in the treatment of gingivitis: a randomised, placebo-controlled clinical trial. Oral Health Prev Dent. 2007;5(4):327-36. PMID 18173095
- [Result] Cohen DW, Friedman LA, Shapiro J, Kyle GC, Franklin S. Diabetes mellitus and periodontal disease: two-year longitudinal observations. I. J Periodontol. 1970 Dec;41(12):709-12. doi: 10.1902/jop.1970.41.12.709. No abstract available. PMID 5275715